CLINICAL TRIAL: NCT01233531
Title: Effects of Cash Transfer for the Prevention of HIV in Young South African Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 068; 11710 (Other: DAIDS ID: 11710); UM1AI068619 (NIH)
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A--Monthly cash transfers (Other): Monthly cash transfer payments
  Interventions: Behavioral: monthly cash transfer payments for attending school
- B--No cash transfers (Other): No cash transfers.
  Interventions: Behavioral: monthly cash transfer payments for attending school; Behavioral: B--No cash transfers

INTERVENTIONS:
Behavioral: monthly cash transfer payments for attending school — In the intervention, young women and their households will be randomized in 1:1 ratio to receive monthly cash transfer payments, conditional on the young woman attending school, or to the control arm. Young women will be recruited at the beginning of grades 8 through 11 in the first year of the study.
Behavioral: B--No cash transfers — No monthly cash transfers
  Arms: B--No cash transfers

SUMMARY:
Cash transfers to young women for staying in school and its effect on acquiring HIV

DETAILED DESCRIPTION:
The overall purpose of this study is to determine whether providing cash transfers to young women and their household, conditional on school attendance, reduces young women's risk of acquiring Human Immunodeficiency Virus (HIV). The overall goal of the Conditional Cash Transfer (CCT) intervention is to reduce structural barriers to education with the goal of increasing school attendance of young women, thereby decreasing their HIV risk.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 13 to 20 years.
* Enrolled in grades 8, 9, 10 or 11 at the beginning of the study at schools in the AHDSS study site
* Intending to continue to live in the study site until the end of the follow-up period.
* Be willing and able to consent/assent to all study procedures including HIV and HSV-2 testing.
* Able to read sufficiently to use ACASI.
* Have a bank or post office account or have documentation to be able to open a bank or post office account (i.e., birth certificate, South African National Identification Book, or passport and proof of residence). Post Office accounts will only be required for participants in the Intervention arm.
* Parent/Legal Guardian who lives with young woman, willing and able to consent to all study procedures including HIV and HSV-2 testing.
* Parent/Legal Guardian has a bank or post office account or has documentation to be able to open a bank or post office account (i.e. South African National Identification Book, or passport and proof of residence). Note that the account may be opened in the name of any adult who resides in the household with the young woman.

Exclusion Criteria:

* Pregnant by self-report at baseline.
* Married at baseline.
* No parent or legal guardian living in household.
* Any other reason that the staff feels would jeopardize the health or well-being of the participant or staff or would prevent proper conduct of the study.

Ages: 13 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2537 (Actual)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
HIV Incidence | 4 years
  To determine whether young women who are randomized to receive CCTs conditional on school attendance have a lower incidence of HIV infection over time compared to young women who are not randomized to receive cash transfers.

SECONDARY OUTCOMES:
HSV-2 incidence | 4 years
  To determine whether young women who are randomized to receive CCTs conditional on school attendance have a lower incidence of Herpes Simplex Virus type 2 (HSV-2) infections over time compared to young women who are not randomized to receive cash transfers.
HSV Incidence | 4 years
  To determine whether young women who receive the CCTs report less unprotected sex, fewer number of sexual partners, younger male partners, an older age of coital debut, a lower incidence of self-reported pregnancy, and greater school attendance compared to young women who do not receive the cash transfers.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Pettifor, Study Chair — University of North Carolina; Xavier Gomez-Olive, Principal Investigator — Wits Rural Public Health and Health Transitions Research Unit; Kathleen Kahn, Principal Investigator — University of Witwatersrand, South Africa; Catherine McPhail, Principal Investigator — Reproductive Health & HIV Research Unit, University of Witwatersrand
Locations (1):
- Agincourt, Acornhoek, South Africa

REFERENCES:
- [Derived] Rosenberg M, Beidelman E, Chen X, Canning D, Kobayashi L, Kahn K, Pettifor A, Kabudula CW. The impact of a randomized cash transfer intervention on mortality of adult household members in rural South Africa, 2011-2022. Soc Sci Med. 2023 May;324:115883. doi: 10.1016/j.socscimed.2023.115883. Epub 2023 Mar 31. PMID 37023659
- [Derived] Jayaweera RT, Goin D, Twine R, Neilands TB, Wagner RG, Lippman SA, Kahn K, Pettifor A, Ahern J. Associations between WASH-related violence and depressive symptoms in adolescent girls and young women in South Africa (HPTN 068): a cross-sectional analysis. BMJ Open. 2022 Jul 5;12(7):e061032. doi: 10.1136/bmjopen-2022-061032. PMID 35790334
- [Derived] DeLong SM, Powers KA, Pence BW, Maman S, Dunkle KL, Selin A, Twine R, Wagner RG, Gomez-Olive FX, MacPhail C, Kahn K, Pettifor A. Longitudinal Trajectories of Physical Intimate Partner Violence Among Adolescent Girls in Rural South Africa: Findings From HPTN 068. J Adolesc Health. 2020 Jul;67(1):69-75. doi: 10.1016/j.jadohealth.2019.12.016. Epub 2020 Feb 13. PMID 32061464
- [Derived] MacPhail C, Khoza N, Selin A, Julien A, Twine R, Wagner RG, Gomez-Olive X, Kahn K, Wang J, Pettifor A. Cash transfers for HIV prevention: what do young women spend it on? Mixed methods findings from HPTN 068. BMC Public Health. 2017 Jul 11;18(1):10. doi: 10.1186/s12889-017-4513-3. PMID 28697762
- [Derived] Pettifor A, MacPhail C, Hughes JP, Selin A, Wang J, Gomez-Olive FX, Eshleman SH, Wagner RG, Mabuza W, Khoza N, Suchindran C, Mokoena I, Twine R, Andrew P, Townley E, Laeyendecker O, Agyei Y, Tollman S, Kahn K. The effect of a conditional cash transfer on HIV incidence in young women in rural South Africa (HPTN 068): a phase 3, randomised controlled trial. Lancet Glob Health. 2016 Dec;4(12):e978-e988. doi: 10.1016/S2214-109X(16)30253-4. Epub 2016 Nov 1. PMID 27815148

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT01233531/Prot_ICF_000.pdf